CLINICAL TRIAL: NCT02810730
Title: Prevalence, With Medical Imaging, of the Parenchymatous and/or Ductal Pancreatic Anomalies of Patients With a 1st Degree Familial History of Pancreatic Adenocarcinoma
Brief Title: Prevalence of Pancreatic Anomalies of Patients With a 1st Degree Familial History of Pancreatic Adenocarcinoma
Acronym: PAPAFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0502198069
Record Dates: First submitted 2016-05-06; First posted 2016-06-23 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Prevalence of Pancreas Adenocarcinomas
Keywords: pancreas; adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Other): Pancreatic MRI in the 6 months following the first consultation
  Interventions: Procedure: Pancreatic MRI

INTERVENTIONS:
Procedure: Pancreatic MRI — Pancreatic MRI in the 6 months following the first consultation

SUMMARY:
Pancreatic adenocarcinoma is the 4th leading cause of cancer in the USA. Its incidence is increasing both in France and in Europe, whereas all the other cancers are decreasing in Europe. Moreover, its seriousness is still high, with a mortality rate higher than the average incidence. The aim of PAPAFA study is to assess the prevalence of the pancreatic anomalies which can be revealed thanks to imaging, for patients having a 1st degree pancreatic adenocarcinoma familial history. This could allow detection of lesions which are less than 10 mm long, and improve the dark prognostic of this pathology.

ELIGIBILITY:
Inclusion Criteria:

* patients with a 1st degree familial history of pancreas adenocarcinoma
* patients older than 40
* patients whose life expectancy is > 3 months
* inform and consent form signed
* patient insured under the French social security system

Exclusion Criteria:

* contraindication to the MRI (pace-maker, implanted metallic material, medical history of allergy to the contrast agent, end-stage renal failure, pregnancy, claustrophobia)
* contraindication to anesthesia to do the echo endoscopy
* 1st degree family history of 2 pancreas adenocarinomas
* medical history of allergy to benzylic alcool
* contraindication to dimeglumine gadobenate
* pregnant or breastfeeding woman, according to the questioning
* subjets who don't have the legal capacity to consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of patients for whom the MRI and/or the echo endoscopy has shown a parenchymatous or ductal pancreatic anomaly | six months after the last inclusion
  For every patients who will have a pancreatic MRI detecting an anomaly, the echo endoscopy will be done. A cytology of the lesion from the echo endoscopy will be done for the solid lesions and for the indetermined cystic lesions (that is to say, the lesions which don't meet the literature set criteria for serous kyst or intraductal papillary and mucinous tumor of the pancreas) ; which is usually done in health care.

SECONDARY OUTCOMES:
Number of patients for whom the MRI has brought to light a parenchymatous and/or ductal pancreatic anomaly | six months after the last inclusion
Number of patients for whom the echo endoscopy has brought to light a parenchymatous and/or ductal pancreatic anomaly | six months after the last inclusion
Height of the lesions | six months after the last inclusion
Correlation between the data from the MRI and those from the echo endoscopy | six months after the last inclusion
Localisation of the lesions | six months after the last inclusion
Number of lesions | six months after the last inclusion
Aspect of the lesion (solid and/or liquid) | six months after the last inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Anne-marie Marion Audibert, Study Director
Locations (9):
- France (9):
  - Clinique Convert, Bourg-en-Bresse
  - Infirmerie Protestante, Caluire-et-Cuire
  - Clinique du Val d'Ouest, Écully
  - Groupe Hospitalier Mutualiste des Eaux Claires, Grenoble
  - Centre des maladies du foie et de l'appareil digestif, Irigny
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Hôpital privé Jean Mermoz, Lyon
  - Clinique des Portes du Sud, Vénissieux
  - Hôpital de Villefranche, Villefranche-sur-Saône